CLINICAL TRIAL: NCT04153058
Title: Randomized Controlled Trials on Clinical Outcomes of Robotic Versus Laparoscopic Assisted Radical Gastrectomy for Advanced Siewert II/III Esophagogastric Junction Adenocarcinoma
Brief Title: Clinical Outcomes of Robotic Versus Laparoscopic Assisted Radical Gastrectomy for Advanced Siewert II/III AEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-018
Record Dates: First submitted 2019-10-20; First posted 2019-11-06 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Esophagogastric Junction Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Assisted AEG Radical Gastrectomy (Experimental): Robotic Assisted Radical Gastrectomy for Advanced Siewert II/III Esophagogastric Junction Adenocarcinoma
  Interventions: Procedure: Robotic Assisted AEG Radical Gastrectomy
- Laparoscopic Assisted AEG Radical Gastrectomy (Active Comparator): Laparoscopic Assisted Radical Gastrectomy for Advanced Siewert II/III Esophagogastric Junction Adenocarcinoma
  Interventions: Procedure: Laparoscopic Assisted AEG Radical Gastrectomy

INTERVENTIONS:
Procedure: Robotic Assisted AEG Radical Gastrectomy — Robotic Assisted Radical Gastrectomy for Advanced Siewert II/III Esophagogastric Junction Adenocarcinoma
  Arms: Robotic Assisted AEG Radical Gastrectomy
Procedure: Laparoscopic Assisted AEG Radical Gastrectomy — Laparoscopic Assisted Radical Gastrectomy for Advanced Siewert II/III Esophagogastric Junction Adenocarcinoma
  Arms: Laparoscopic Assisted AEG Radical Gastrectomy

SUMMARY:
The purpose of this study is to explore the clinical outcomes of the robotic assisted radical gastrectomy for advanced Siewert II/III esophagogastric junction adenocarcinoma（cT2-4a, N-/+, M0）

DETAILED DESCRIPTION:
In recent years, the incidence of gastric cancer has been decreasing year by year in the world, but the incidence of adenocarcinoma of the esophagogastric junction (AEG) has shown a significant upward trend, especially in Western countries such as Europe and the United States. The prognosis of AEG is poor, therefore, it is extremely necessary to establish AEG's best diagnosis and treatment strategies to improve the long-term outcome of AEG. Robotic surgery has been developed with the aim of improving surgical quality and overcoming the limitations of conventional laparoscopy in the performance of complex mini-invasive procedures. The study is designed to explore the clinical outcomes of the robotic assisted radical gastrectomy for advanced Siewert II/III esophagogastric junction adenocarcinoma (cT2-4a, N-/+, M0) by comparing with laparoscopic assisted.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT2-4a(clinical stage tumor), N-/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
* Expected to perform total gastrectomy with D2+No.19+No.20 lymph node dissction to obtain R0 resection sugicall results.
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) class I to III
* Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastric surgery (except ESD/EMR (Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection )for gastric cancer)
* Gastric multiple primary carcinoma
* Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging
* History of other malignant disease within the past 5 years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within the past 6 months
* History of cerebrovascular accident within the past 6 months
* History of continuous systematic administration of corticosteroids within 1 month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of the predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months
  3-year disease free survival rate

SECONDARY OUTCOMES:
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year recurrence pattern | 36 months
  3-year recurrence pattern
overall postoperative morbidity rates | 30 days
  overall postoperative morbidity rates
intraoperative morbidity rates | 1 day
  intraoperative morbidity rates
overall postoperative serious morbidity rates | 30 days
  overall postoperative serious morbidity rates
number of retrieved lymph nodes | 14 days
  number of retrieved lymph nodes
Time to first ambulation | 30 days
  Time to first ambulation is used to access the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus is used to access the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet is used to access the postoperative recovery course.
Time to soft diet | 30 days
  Time to soft diet is used to access the postoperative recovery course.
Duration of hospital stay | 30 days
  Duration of hospital stay is used to access the postoperative recovery course.
The amount of abdominal drainageare | 30 days
  The amount of abdominal drainageare is used to access the postoperative recovery course.
postoperative nutritional status | 3, 6, 9 and 12 months
  Weight and height will be combined to report BMI in kg/m^2. The variation of BMI in kg/m^2 on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status.
Hospitalization costs | 30 days
  Hospitalization costs

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No